CLINICAL TRIAL: NCT01456910
Title: Evaluation and Effects of a Resistance Training Program and Its Relationship With the Labor Inclusion of the Disabled Intellectual
Brief Title: Resistance Training Program, Labor Inclusion, Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Andrea Glaucy Davim Raulino, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0018.0.012.000-09
Record Dates: First submitted 2011-10-14; First posted 2011-10-21 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Mental Retardation; Body Composition, Beneficial; Muscle Weakness
Keywords: Physical education; People with mental disabilities; muscular strength dynamometer; Performance Evaluation; Occupational health
MeSH Terms: conditions — Intellectual Disability; Glucocorticoid Receptor Deficiency; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working group (Experimental): G1 intervention group of 20 participants aged 14-36 years old and mild to severe intellectual disability of both gender.
  Interventions: Behavioral: Resistance Training Program
- Daily Living (Active Comparator): G2 control group continue usual routine
  Interventions: Behavioral: Resistance Training Program

INTERVENTIONS:
Behavioral: Resistance Training Program — Frequency, volume, repetitions, load, interval
  Other Names: Biodex-System3Pro® dynamometer; Activities of Daily Living adapted to work productivity; InBody 720

SUMMARY:
Resistance exercise (RE) has been proposed as a possible strategy for prevention and rehabilitation of diseases. The increase in both muscle strength and the ability to perform tasks of day-to-day work environment and are well-characterized benefits of this type of training. The literature has been investigating the effectiveness of the RE for humans, yet few studies have been conducted with intellectual disabilities (ID). It is known that a sedentary lifestyle contributes to the development of cardiovascular disease, type 2 diabetes, hypertension, arthritis, and stress, depression, difficulty in socializing, stigma and discrimination. In particular, the ID is less active and is more likely to develop secondary diseases.

DETAILED DESCRIPTION:
This study aimed to correlate peak torque with work task performance (WTP) after application of resistance training program (RTP), consisting of 40 sessions, twice a week lasting 90 minutes each session. The sample was constituted by 40 individuals, which were selected from a survey of the records filed at Parents and Friends of Exceptional Children of Federal District/Brazil Association (APAE/DF), taking into consideration the following criteria: be inserted in the Professional Education and Labor Program (PELP) of APAE/DF, age between 14 and 36 years for being the most active labor, show no physical disabilities, do not have cardiac problems, who wish to inform the study and voluntarily sign the Free and Informed Term of Consent with their tutors. Although the participants are residents of various cities in the Federal District, it was not possible to avoid selection bias, since the sample was selected from a single institution, limiting, thus, generalization of results.

After performing the pre-testing peak torque, by Biodex System3Pro Dynamometer, and WTP through 800m, climbing stairs and labor skill (to decorate two tables for 4 people, separated by one meter, for lunch with 2 tablecloths, 8 plates, 8 forks, 8 knives and 8 glasses), participants were randomly assigned to experimental groups - G1 (20 participants) and control - G2 (20 participants), and matched according to age, sex and per capita income, in order to form groups with similar characteristics. The G1 group participated in the RTP in number of eight, four for the upper limbs and four for the lower limbs. In order to avoid confounding bias, participants in the G2 group, along with their tutors, were instructed to continue with their daily activities normally and did not participate in RTP, as well as the G1 also instructed not to participate in other physical activities.

The first Monthly cycle (two weeks) was developed in order to familiarize participants with the equipment and learn how to perform the exercises, avoiding, thus, evaluation bias. Subsequently, we applied the test of one maximum repetition - 1MR, to elaborate a spreadsheet on individual training with the participants. The second, third and fourth Monthly cycles were developed according to the spreadsheet elaborated timeline and orientation of the instructors, which were duly informed. After four months of intervention, all 40 participants were reassessed.

This study was approved by the Ethics and Research Committee at the University of Brasilia under the resolution 196/96 of the National Health Ministry of Health with the record 21/09 and is registered in the National Information System on Ethics in Research Involving Human Subjects - SISNEP with the number of Certificate of Presentation for Ethics Appreciation - CAAE: 0018.0.012.000-09.

The Institutions Association of Parents and Friends of Exceptional Children of Federal District, Resistance Exercise Laboratory of the Faculty of Physical Education at the University of Brasilia, Physics Resistance Gym and Nutriment - Center of Medicine Nutrition were contacted and informed about the research procedures by requesting formal practice of testing due to the participants in this study by signing the Declaration of Institutional Science.

ELIGIBILITY:
Inclusion Criteria:

1. Be intellectually disabled
2. Be aged between 16 and 36 years
3. Understand the information provided by the researcher during data collection with the isokinetic dynamometer
4. Understand the information provided by the researcher during the course of the program of resistance exercise
5. Do not report pain in the joint tested
6. Do not have limitations in range of motion of the knee joint
7. Do not be swollen in the joint
8. Interest in participating in the study
9. Sign the Statement of Consent or your parent.

Exclusion Criteria:

1. Provide cognitive impairment such that he does not understand the instructions necessary to collect data regarding the strength of knee flexion-extension with the isokinetic dynamometer
2. Cognitive impairment such that he does not understand the instructions needed to perform the necessary movements of resistance exercise program
3. Display heart
4. Report pain before the test
5. Present joint swelling
6. Use a pacemaker or other electromedical equipment
7. Failure to properly hold the electrodes
8. Do not have an interest in participating in the study;
9. Not having signed an informed consent or your parent.

Ages: 14 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea GD Raulino, MD, Principal Investigator — University of Brasilia
Locations (2):
- Brazil (2):
  - Association of Parents and Friends of Exceptional Children of Federal District/Brazil; Resistance Exercise Laboratory of the Faculty of Physical Education at the UnB/Brazil; Physics Resistance Gym and Nutrimed Clinics - Center of Medicine Nutrition, Brasília, Federal District
  - University of Brasília, Brasília, Federal District

REFERENCES:
- [Result] Stopka C, Limper L, Siders R, Graves J, Goodeman A, Silvestone E. Effects of a supervised resistence training program on adolescents and young adults with mental retardation. J Strength Cond Res 1994; 8(3): 184-7. Croce RV, Horvat M. Effects of reinforcement-based exercise on fitness and work productivity in adults with mental retardation. Adapt Phys Activ Q 1992; 9:148-78. Shields N, Taylor NF, Dodd KJ. Effects of a community-based progressive resistance training program on muscle performance and physical function in adults with Down syndrome: a randomize controlled trail. Arch. Phys. Med. Rehabil 2008; 89: 1215-20. Zetts R, Horvat M, Langone J. Effects of a community-based progressive resistence training program the work productivity of adolescents with moderate to severe intellectual disabilities. Educ Train Ment Retard 1995; 30:166-78. Smail K, Horvat M. Relationship of muscular strength on work performance in high school students with mental retardation. Educ. Train Dev. Disabil. 2006 Dec; 41(4):410-19. Andreotti RA, Okuma SS. Validação de uma bateria de testes de atividades da vida diária para idosos fisicamente independentes. Rev paul educ fís 1999; 13(1):46-66. Carmeli E, Ayalon M, Barchard S, Sheklow SL, Reznik AZ. Isokinetic leg strength of institutionalized older adults with mental retardation with and without Down's syndrome. J Strength Cond Res 2001; 16(2): 316-20. Rimmer JH, Kelly LE. Effects of a resistance training program of adults with mental retardation. Adapt Phys Activ Q 1991; 8:146-53. Mendoca GV, Pereira FD, Fernhall B. Effects of combined aerobic and resistence exercise training in adults with and without Down syndorme. Arch Phys Med Rehabil 2011; 92: 37-45. Shields N, Taylor NF, Fernhall B. A study protocol of randomized controlled trial to investigate if a community based strength training programme improves work task performance in young adults with Down syndrome. BMC Pediatr 2010; 10-17.
- See also: National information on ethics in research involving human — http://portal2.saude.gov.br/sisnep/pesquisador/Projetos_Aprovados.cfm?uf=DF&inicio=01/01/2009&fim=01/01/2010